CLINICAL TRIAL: NCT06751030
Title: Community, Home-based Education, Screening Services (CHESS) Strategy to Increase Cervical Cancer Control Access for HIV-Positive Women in Nigeria
Brief Title: Community, Home-based Education, Screening Services Strategy to Increase Cervical Cancer Control Access for HIV-Positive Women in Nigeria
Status: Recruiting | Type: Observational
Sponsor: Emory University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Lisa Flowers, Professor, Emory University
Other Study IDs: STUDY00004817; U01CA275113 (NIH)
Record Dates: First submitted 2024-12-20; First posted 2024-12-27 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: HIV; Cervical Cancer
Keywords: Women Living With HIV; cervical cancer screening
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Women living with HIV: During the screening process:
  * Women testing negative for high-risk HPV (HrHPV) will complete participation one year after their test results, at which time they will be invited to retest.
  * Women living with HIV (WLWH) testing positive for HrHPV will have endpoints based on treatment outcomes:
    * Other HrHPV types (not 16/18/45):
      * Endpoint: One year post-VIA (visual inspection with acetic acid).
      * VIA-positive patients will receive thermal ablation treatment.
      * VIA-negative patients will have repeat VIA or standard screening after one year.
    * HrHPV types 16/18/45:
      * Endpoint: Two years post-treatment.
      * Follow-up includes repeat HPV self-collection, VIA, biopsies, and further treatment (thermal ablation or excision) if needed.
  WLWH testing positive for HrHPV 16/18/45 via self-collection will be notified by a Mentor Mother, who, along with Nigerian clinical staff, will assist in scheduling VIA. Treatment follows the standard of care protocol.
  Interventions: Behavioral: The Mother Mentor program; Diagnostic Test: GeneXpert HPV test

INTERVENTIONS:
Behavioral: The Mother Mentor program — The MOther MENTor (MoMent) program in Nigeria pairs trained treatment-experienced Women living with HIV (WLWH), known as Mentor Mothers (MMs), with new mothers who are newly diagnosed with HIV to improve access to and retention in HIV care
  Other Names: MoMent Program
Diagnostic Test: GeneXpert HPV test — A cervical cancer screening tool.

SUMMARY:
The goal of this observational study is to focus on adapting and implementing a program to promote HPV and cervical cancer (CC) screening and follow-up treatment for HIV-positive women, with three specific aims:

* Adaptation: Use stakeholder deliberation to tailor the successful MoMent program for this population.
* Implementation and Assessment: Deploy the adapted MoMent program and evaluate its reach, effectiveness, adoption, and fidelity.
* Evaluation: Conduct a post-implementation process evaluation to identify barriers and facilitators to the program's maintenance and sustainability.

DETAILED DESCRIPTION:
Despite the increased risk of cervical cancer (CC) among women living with HIV (WLWH), access to CC screening in Nigeria remains limited. While advances in prevention programs and antiretroviral therapy have reduced other AIDS-associated malignancies, CC risk in WLWH persists. This study aims to leverage Nigeria's existing HIV treatment infrastructure to integrate home-based CC (HCC) screening for WLWH.

The approach involves adapting the MoMent (MOther MENTor) peer-based HIV support program to include HCC screening and evaluating its implementation and sustainability using the Consolidated Framework for Implementation Research (CFIR) and RE-AIM frameworks. The study has three key aims:

* Adapting the MoMent program to promote home-based HPV screening and follow-up treatment through stakeholder deliberation.
* Implementing and assessing the program's reach, effectiveness, adoption, and fidelity with a sample of 1,500 WLWH.
* Conducting a post-implementation evaluation to identify barriers and enablers for program maintenance and scalability.

Stakeholder input, including perspectives from WLWH, peer counselors, clinical managers, and policymakers, will guide the program's design and execution. By integrating stakeholder insights and addressing systemic challenges, the study aims to advance CC control in Nigeria and provide a scalable model for implementing cancer control strategies for people living with HIV in low- and middle-income countries globally.

ELIGIBILITY:
Inclusion Criteria:

- Patients must be able to perform vaginal self-collection as well as give informed consent

Exclusion Criteria:

* Male gender
* Age <25 or >50
* Unknown or negative HIV status
* Pregnancy
* Hysterectomy
* Inability to give informed consent Inability/refusal to perform vaginal self-collection

Ages: 25 Years to 50 Years | Sex: Female
Age Groups: Adult
Study Population: Aim 1: The stakeholder deliberation conferences will include stakeholders from the following groups:
  * State and National Policymakers
  * Organizational-clinical managers
  * Mentor mothers
  * Women living with HIV (WLWH) Since this is a socio-behavioral component, pregnant individuals may partake. All individuals who take part in this portion of the study will be above 18 and capable of providing informed consent.
  Aim 2: This study will only include WLWH aged 25-50. Pregnant individuals will not be included due to the potential for treatment of precancerous lesions. All individuals who partake in the study will be older than 18 and capable of providing informed consent.
Sampling Method: Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2024-12-03 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Program Reach | Baseline, Month 6, Month 18
  Reach evaluated through the provision of home test kits to eligible women, returned samples, number of WLWH positive for high-risk HPV (hrHPV) treated, persistence or reoccurrence of hrHPV or cervical precancerous lesions post-treatment, and correlation of these results with CD4 and HIV viral load.
Effectiveness of the Program | Baseline, Month 6, Month 18
  Effectiveness evaluated through the provision of home test kits to eligible women, returned samples, number of WLWH positive for high-risk HPV (hrHPV) treated, persistence or recurrence of hrHPV or cervical precancerous lesions post-treatment, and correlation of these results with CD4 and HIV viral load.
Adoption of the program | Baseline, Month 6, Month 18
  Adoption will be measured through the proportions of MMs who complete training and WLWH who return self-collected (SC) samples
Fidelity of the program | Baseline, Month 6, Month 18
  Will be measured by peer leaders' monitoring of practices, as well as measuring system barriers and added MoMent program costs per completed home screening

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Flowers, MD, MPH, Principal Investigator — Emory University
Locations (3):
- Nigeria (3):
  - APIN Health Initiatives, Abuja
  - University of Ibadan, Ibadan
  - Nigeria Institute of Medical Research (NIMR, Lagos

IPD SHARING:
Plan to Share IPD: Yes
Data shared:
  De-identified sociodemographic data (e.g., race/ethnicity, age). Health behavior and health care utilization data from medical records. Cervical pathology results, HPV testing data, laboratory tests (e.g., CD4 and viral load), prescribed HIV medications, and adherence data.
  Qualitative data from in-depth interviews and focus group discussions, coded and anonymized.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Start Date: After primary analyses have been completed and results are published (expected within 12 months of study completion).
  End Date: Indefinitely, contingent on adherence to data-sharing agreements
Access Criteria: Researchers will submit a Data Analysis Request Form, detailing their proposed analysis, purpose, and data needed.
  Data access will be granted following review and approval. Approved users will sign a Data Use and Confidentiality Agreement. Anonymized data will be shared securely via a designated data repository or encrypted file transfer.
  Researchers must commit to using the data for specified purposes, implementing secure data storage, and destroying or returning the data after analyses are completed.

REFERENCES:
- [Derived] Ogunsola O, Gaydos LM, Ajayi O, Dieci M, Kaonga N, Awolude O, Ezemelue P, Staple T, Salami K, Idigbe I, Ezechi O, Flowers L. The CHESS Protocol: A Mixed-Methods Evaluation of an HPV Screening Intervention for Women Living With HIV in Nigeria. Int J Public Health. 2025 Aug 14;70:1608716. doi: 10.3389/ijph.2025.1608716. eCollection 2025. PMID 40895387